CLINICAL TRIAL: NCT03180112
Title: The Association Between Herpes Simplex Viruses (Type One and Two) and Autism Spectrum Disorders
Brief Title: The Association Between Herpes Simplex Viruses and Autism
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khalaf A Sayed, principle investigator, Assiut University
Other Study IDs: HA
Record Dates: First submitted 2017-06-01; First posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Enzyme-Linked Immunosorbent Assay; Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — quantitative polymerase chain reaction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: Children suffering from Autism Spectrum disorders of variable grades attending to assiut University Children Hospital aged between six months and five years.
  Interventions: Genetic: enzyme linked immunosorbent assay and polymerase chain reaction
- control group: Healthy children of matching age and sex.
  Interventions: Genetic: enzyme linked immunosorbent assay and polymerase chain reaction

INTERVENTIONS:
Genetic: enzyme linked immunosorbent assay and polymerase chain reaction — Blood samples will be collected and analyzed for herpes simplex viruses (type one and two) antibody by sensitive enzyme-linked immunosorbent assay and quantitative polymerase chain reaction.

SUMMARY:
Autism spectrum disorders are pervasive developmental disorders that include autistic disorder, Asperger's disorder, and pervasive developmental disorder-not otherwise specified.They are characterized by stereotypic behaviors, variable deficits in language and social skills and a wide range of other behavioral problems. Autism spectrum disorders manifest during childhood and at least thirty percent present with sudden clinical regression of development around three years of age.

DETAILED DESCRIPTION:
Over the last twenty years, there has been an impressive rise in Autism spectrum disorders with current prevalence estimates being about one over one hundred children.

Herpes simplex virus encephalitis is the leading cause of sporadic, nonepidemic encephalitis in children and adults in the United States. It is an acute necrotizing infection generally involving the frontal and/or temporal cortex and the limbic system and, beyond the neonatal period, is almost always caused by Herpes simplex virus type on.

The etiology of autism is unknown; data suggest that autism results from multiple etiologies with both genetic and environmental contributions. One proposed etiology for autism is viral infection very early in development. The mechanism, by which viral infection may lead to autism, be it through direct infection of the central nervous system, through infection elsewhere in the body acting as a trigger for disease in the central nervous system, through alteration of the immune response of the mother or offspring, or through a combination of these, is not yet known.

Many encephalitic patients had temporal lobe involvement. Autism results from neuropathology relating to the temporal lobes. They speculate the differences in the extent and neuropathologies of the temporal lobes contribute to the heterogeneity of autism. Also, herpes viruses can induce a variety of proinflammatory cytokines during infections, along with elevated interferon in the brain during Herpes simplex virus encephalitis.

ELIGIBILITY:
Inclusion Criteria:

1. Children suffering from Autism spectrum disorders.
2. Age between six months and five years

Exclusion Criteria:

1. Genetic disorders.
2. History of metabolic or neurodegenerative disease.
3. Gross motor delay.
4. Audiologic problems.
5. Mental retardation.
6. Other psychiatric problems.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children suffering from Autism Spectrum disorders of variable grades attending to Assuit University Children Hospital and the same number of healthy children of matching age and sex as a control.
  Age between six months and five years
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2018-08-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
relationship between herpes simplex viruses infections and development of autism. | 12 month
  Detection of herpes simplex viruses antibody titre by sensitive enzyme linked immunosorbent assay and detection of herpes simplex viruses titre by quantitative polymerase chain reaction

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson CP, Myers SM; American Academy of Pediatrics Council on Children With Disabilities. Identification and evaluation of children with autism spectrum disorders. Pediatrics. 2007 Nov;120(5):1183-215. doi: 10.1542/peds.2007-2361. Epub 2007 Oct 29. PMID 17967920
- [Background] Zappella M. Autistic regression with and without EEG abnormalities followed by favourable outcome. Brain Dev. 2010 Oct;32(9):739-45. doi: 10.1016/j.braindev.2010.05.004. Epub 2010 Aug 12. PMID 20708360
- [Background] Fombonne E. Epidemiology of pervasive developmental disorders. Pediatr Res. 2009 Jun;65(6):591-8. doi: 10.1203/PDR.0b013e31819e7203. PMID 19218885
- [Background] Libbey JE, Sweeten TL, McMahon WM, Fujinami RS. Autistic disorder and viral infections. J Neurovirol. 2005 Feb;11(1):1-10. doi: 10.1080/13550280590900553. PMID 15804954
- [Background] DeLong GR, Bean SC, Brown FR 3rd. Acquired reversible autistic syndrome in acute encephalopathic illness in children. Arch Neurol. 1981 Mar;38(3):191-4. doi: 10.1001/archneur.1981.00510030085013. PMID 6162440
- [Background] Gillberg C. Onset at age 14 of a typical autistic syndrome. A case report of a girl with herpes simplex encephalitis. J Autism Dev Disord. 1986 Sep;16(3):369-75. doi: 10.1007/BF01531665. No abstract available. PMID 3558293
- [Background] Ghaziuddin M, Tsai LY, Eilers L, Ghaziuddin N. Brief report: autism and herpes simplex encephalitis. J Autism Dev Disord. 1992 Mar;22(1):107-13. doi: 10.1007/BF01046406. No abstract available. PMID 1592760
- [Background] Hetzler BE, Griffin JL. Infantile autism and the temporal lobe of the brain. J Autism Dev Disord. 1981 Sep;11(3):317-30. doi: 10.1007/BF01531514. PMID 6189814
- [Background] Dalod M, Salazar-Mather TP, Malmgaard L, Lewis C, Asselin-Paturel C, Briere F, Trinchieri G, Biron CA. Interferon alpha/beta and interleukin 12 responses to viral infections: pathways regulating dendritic cell cytokine expression in vivo. J Exp Med. 2002 Feb 18;195(4):517-28. doi: 10.1084/jem.20011672. PMID 11854364
- [Background] Salazar-Mather TP, Hamilton TA, Biron CA. A chemokine-to-cytokine-to-chemokine cascade critical in antiviral defense. J Clin Invest. 2000 Apr;105(7):985-93. doi: 10.1172/JCI9232. PMID 10749577
- [Background] Legaspi RC, Gatmaitan B, Bailey EJ, Lerner AM. Interferon in biopsy and autopsy specimens of brain. Its presence in herpes simplex virus encephalitis. Arch Neurol. 1980 Feb;37(2):76-9. doi: 10.1001/archneur.1980.00500510034004. PMID 7356411